CLINICAL TRIAL: NCT03688685
Title: A Phase 2a Open-Label Study to Evaluate the Safety, Tolerability and Efficacy of CAD-1883 Oral Treatment in Adults With Essential Tremor
Brief Title: A Clinical Study to Evaluate CAD-1883 in Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cadent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAD1883-201
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Essential Tremor
Keywords: ET; Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label study of CAD-1883 (Experimental): Open-label study designed to evaluate the safety, tolerability, and efficacy of CAD-1883 administered twice daily orally to adult subjects with ET
  Interventions: Drug: CAD-1883

INTERVENTIONS:
Drug: CAD-1883 — Treatment groups receiving twice-daily oral dosing of CAD-1883 for a treatment period of 14 days.

SUMMARY:
This is an open-label study designed to evaluate the safety, tolerability and efficacy of CAD-1883, a positive allosteric modulator of the SK channel, administered twice daily orally to adult patients with ET. Patients with the diagnosis of ET based on the Movement Disorder Society (MDS) criteria with a documented severity of tremor based on the clinician-administered TETRAS Performance Subscale are eligible to be enrolled in the study.

DETAILED DESCRIPTION:
This is an open-label study designed to evaluate the safety, tolerability and efficacy of CAD-1883, a positive allosteric modulator (PAM) of the SK channel, administered twice daily orally to adult subjects with ET. Positive modulation of the small-conductance calcium-activated potassium channels (SK) present in different regions of the brain aims to increase the channel sensitivity to calcium resulting in reduction in neuronal firing rate. In patients with ET, improving the regularity of firing of action potentials in the olivo-cerebellar network can lead to improvement in motor function.

During the Screening period, each subject will undergo full assessment including medical and treatment history for ET, physical examination and other screening assessments. Patients with the diagnosis of ET based on the Movement Disorder Society (MDS) criteria with a documented severity of tremor based on the clinician-administered TETRAS Performance Subscale are eligible to be enrolled in the study. The study consists of treatment groups receiving twice daily oral dosing of CAD-1883 for a treatment period of 14 days.

This study is designed to enable the assessment of safety and tolerability of CAD-1883 in patients with ET as well as the determination of early treatment effect on reducing the magnitude and severity of tremor while limiting the potential risk associated with a novel investigational drug.

Safety and tolerability will be monitored throughout the study duration including in-clinic assessments of adverse events (AEs), serious adverse events (SAEs), vital signs, 12-lead ECG, urinalysis, hematology, clinical chemistry, and CAD-1883 plasma concentration level on Days 1, 7, 14 and 21.

Efficacy will be evaluated using the clinician-administered TETRAS Performance Subscale as well as the use of a wearable sensor in the clinic and at home.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged between 18 and 75 years old, inclusive, with history of tremor that fulfills the diagnostic criteria of ET according to Movement Disorder Society (MDS) Consensus Statement on the classification of tremors from the task force on tremor of the International Parkinson and Movement Disorder Society (Bhatia, 2018).
2. Duration of ET illness since the first symptoms were noticeable of at least 3 years or more prior to screening, based on the subject's self-report, with onset prior to age 65 years old, per the Principal Investigator's assessment during screening.
3. Except for ET, subjects must be otherwise healthy as determined by the Investigator, based upon a medical evaluation including medical history, physical examination, laboratory tests, and 12-lead ECG.
4. Subjects are able to understand study activities required, can give written informed consent, and are willing to comply with the requirements and restrictions of the study.
5. Women of childbearing potential must undertake a pregnancy test with documented negative serum pregnancy test at Screening and negative urine pregnancy test result at Pre-dose, Days 7 and 14 before administration of the study drug, and then at the Follow-up visit (Day 21).
6. Postmenopausal women must have had ≥365 days of spontaneous amenorrhea, with documented follicle-stimulating hormone (FSH) ≥38 IU/mL, prior to screening. If needed, per Investigator's judgment, FSH level can be performed at Screening.
7. Surgically sterile women must have documentation of a hysterectomy, bilateral ovariectomy, or bilateral tubal ligation.
8. Female subjects with reproductive potential and male subjects with reproductive potential or who have female partners of reproductive potential, must agree to use two effective methods of contraception from signing informed consent until 90 days after the last dose of study drug. Acceptable forms of contraception include double barrier (ie, condom with spermicide); surgically sterilized partner (180-day minimum); or abstinence.

Exclusion Criteria:

1. Prior or ongoing medical condition or any abnormal finding on the Screening visit physical exam, ECG, laboratory testing that, in the Investigator's opinion, could adversely affect the safety of the subject or the conduct of the study assessments.
2. Any neurological abnormality other than ET upon neurological exam, including dystonia, ataxia, or any other neurodegenerative disease, including multiple sclerosis or Parkinson's disease.
3. Significant cognitive impairment or dementia that, in the opinion of the Investigator, would interfere with participation in the study.
4. An unstable thyroid condition that, per the Investigator's judgment, has not stabilized over the past 90 days prior to screening. This includes current clinical history of hypo- or hyperthyroidism, thyrotoxicosis or significant abnormality of thyroid function testing at Screening.
5. History of, or evidence of psychogenic tremor at Screening.
6. History of anaphylaxis, hypersensitivity reactions (including to any of CAD-1883 excipients), or clinically significant drug allergies.
7. Alkaline phosphatase, aspartate aminotransferase (AST), and/or alanine aminotransferase (ALT) level >2.0 x upper limit of normal (ULN) at Screening and/or at Pre-dose.
8. Serum creatinine >120 μmol/L and/or creatinine clearance <60 mL/min (according to Cockcroft-Gault formula) at Screening and/or at Pre-dose.
9. Total bilirubin >2.0 x ULN at Screening and/or at Pre-dose. Note: isolated bilirubin >2.0 x ULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%.
10. History of Long QT syndrome and/or QTcF (Fridericia's correction) interval >450 msec (males) or >470 msec (females) per 12-lead ECG done at Screening.
11. History of Alcohol Use Disorder per Diagnostic Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria.
12. History of human immunodeficiency virus (HIV) infection or positive screening result for: HIV 1 or 2 antibodies, hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb), or hepatitis C virus antibody (HCVAb).
13. Has a diagnosis of epilepsy or any history of seizure as an adult, head trauma, stroke, transient ischemic attack within 1 year prior to Screening, unexplained loss of consciousness within 1 year prior to Screening, or any lifetime history of asymptomatic or symptomatic orthostatic hypotension (eg, postural syncope).
14. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class 3 or 4), or clinically significant conduction abnormalities (eg, unstable atrial fibrillation) within 1 year prior to screening.
15. Any major psychiatric disorder that is uncontrolled (for the past 90 days) that, per the Investigator's judgment, can interfere with any of the study procedures.
16. Subject has cancer, except for the following: basal cell carcinoma or successfully treated squamous cell carcinoma of the skin; cervical carcinoma in situ; prostatic carcinoma in situ; or other malignancies curatively treated and with no evidence of disease recurrence for at least 3 years.
17. Subjects with scheduled surgeries during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-23 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Cadent Investigational Site, Anniston, Alabama
  - Cadent Investigational Site, Rogers, Arkansas
  - Cadent Investigational Site, San Diego, California
  - Cadent Investigational Site, Hallandale, Florida
  - Cadent Investigational Site, Farmington Hills, Michigan
  - Cadent Investigational Site, St Louis, Missouri
  - Cadent Investigational Site, Dayton, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open-label Study of CAD-1883
Started | 25
Completed | 21
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Study of CAD-1883
Number analyzed (Participants) | 25
Age, Continuous [Median (Standard Deviation); unit: years] | 67 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Occurrence and Severity of Treatment Emergent AEs.
Description: Number of subjects who experienced TEAEs and the severity of those TEAEs.
Time Frame: Time of signed informed consent until 21 days after first treatment
Measure: Number; unit: participants
Arm/Group | Open-label Study of CAD-1883
Number analyzed (Participants) | 25
participants
  Subjects with at least 1 TAE | 13
  Subjects with Mild AE | 9
  Subjects with Moderate AE | 2
  Subjects with Severe AE | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time the subject signed the informed consent form until the Follow-Up Visit at Day 21.
Arm/Group | Open-label Study of CAD-1883
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label Study of CAD-1883 (N=25)
Fatigue (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor must review results communications prior to public release and can embargo communications regarding trial results. At least sixty (60) days prior to submission for publication or presentation, Institution or Investigator shall submit in writing to sponsor for review or comment of any proposed oral or written publication. The sponsor can require changes to the communication and can delay the publication an additional sixty (60) days.

DOCUMENTS (2):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03688685/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/85/NCT03688685/SAP_001.pdf